CLINICAL TRIAL: NCT04131946
Title: Assessing the Effectiveness of a Community-Based Colorectal Cancer Screening Intervention
Brief Title: Cancer Screening; Access; Awareness; Navigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Karriem S. Watson, Principal Investigator, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2019-0920
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer Screening

STUDY DESIGN:
Intervention Model Description: Experimental and Standard of care arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Intervention Group/Arm 1 (Experimental): Community navigators will work with local businesses (barber shop, hair salon) to identify and screen eligible community members within or near the South Shore community area. The navigator will engage with each potential participant using the attached script. If the participant is interested, the navigator will document the participant's contact information, and assist the participant in obtaining and returning their FIT.
  Community navigators will attend community events to post the informational flyer and provide education about CRC to community members. At these events, they will identify and screen eligible community members within or near the South Shore community area. The navigator will engage with each potential participant using the attached script. If the participant is interested, the navigator will document the participant's contact information, and assist the participant in obtaining and returning their FIT.
  Interventions: Other: Community-Based (Intervention Arm)
- Standard of Care (Control) Arm 2 (No Intervention): These procedures are a detailed summary of the existing lay navigation program at Mile Square Health Center (MSHC). These procedures are unrelated to our research, except to demonstrate how the existing navigation program from which we will obtain deidentified data works.
  Lay clinic navigator use clinic schedules and walk-ins to identify and screen eligible participants within the Englewood MSHC. The navigator engages with each potential participant using standard scripted language. For interested patients, the navigator documents interest and FIT dispensing as appropriate, and assists the patient in obtaining and returning their FIT.
  Lay clinic navigators attend community events as normally scheduled to provide community-based health education and referral to the MSHC. At these events, they identify and screen eligible community members within the Englewood community area.

INTERVENTIONS:
Other: Community-Based (Intervention Arm) — Community dispensed FIT
  Arms: Community Intervention Group/Arm 1

SUMMARY:
To assess the feasibility and efficacy of community-based Colorectal Cancer (CRC) screening intervention in increasing CRC screening rates To evaluate individual-level knowledge related to CRC screening and risk factors To characterize individual -level facilitators and barriers to engaging in CRC screening and related diagnostic tests and treatment when applicable.

DETAILED DESCRIPTION:
To address the multiple determinants of health that impact CRC screening in the South Shore community in the University of Illinois Cancer Center's catchment area by conducting an experimental intervention to test the effectiveness of Fecal immunochemical test (FIT) tests dispensed by community stakeholders (community-dispensed) versus FIT tests dispensed using standard of care procedures by a clinic dispensed FIT test return rates. This study will follow American Cancer Society (ACS) guidelines for FIT testing, with the South Shore community area assigned to the intervention group (community-dispensed). CRC screening within the Mile Square Englewood Health Center, using standard of care, will serve as our control group to use for comparison (clinic-dispensed). The intervention will include a multifaceted approach to health education and community engagement focused on CRC led by a team of trusted health champions (community leaders, a barber, a hair salon, and community health workers) in the South Shore community area.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 45-74
* Speaks English and resides in or near the South Shore community area or utilizes the Mile Square Englewood Heath Center
* Have not had CRC screening in the previous 12 months

Exclusion Criteria:

* Adults ages <45 or >75
* Does not speak English
* Does not reside in or near the South Shore Community area and do not utilize Mile Square Englewood Heath Center
* Have had CRC screening in the previous 12 months

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility and efficacy of conducting a community-based CRC screening intervention in increasing CRC screening rates | 3 years
  Evaluate feasibility and efficacy of conducting a community-based navigation program for CRC screening. In both arms of the study, we will examine the number of participants provided with health education about colorectal cancer, number of FITs distributed, and number of FITs returned. We will summarize the number of persons screened positive and negative, and determine the proportion of positive screening who are referred to clinical care, and at the Mile Square South Shore and Englewood sites through our community navigation program (intervention) and existing MSHC lay clinical navigation program. We will compare the FIT return rate and average return time at the South Shore and Englewood sites to determine if the rates and times are similar. We will also determine return rates and times for participants who screen positive and are navigated to return the MSHC for diagnostic testing, and make comparisons across the intervention and control arms
Evaluate individual-level knowledge related to CRC screening and risk factors | 3 years
  Assess knowledge related to CRC screening and risk factors as measured by our short survey that participants will return with their FIT. We will summarize the frequency and percentage of respondents who have had a prior CRC screening, in addition to the frequency and percentage of respondents who select the correct answers on knowledge questions.
Characterize individual -level facilitators and barriers to engaging in CRC screening and related diagnostic tests and treatment when applicable | 3 years
  Evaluate facilitators and barriers people living in or near the South Shore communities experience related to CRC screening and related follow-up. We will summarize the respondent responses to survey questions about barriers and facilitators

CONTACTS AND LOCATIONS:
Overall Officials: Karriem S Watson, DHSc, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - University of Illinois, Chicago, Illinois
  - Mile Square Health Center - Englewood, Chicago, Illinois

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT04131946/Prot_SAP_000.pdf